CLINICAL TRIAL: NCT07025434
Title: Effects of Hip Bump Manipulation Versus Sham Treatment on Hip Internal Rotation, External Rotator Strength, and Bipodal Landing in Healthy Adults Aged 18-45: A Single-Blinded Randomized Controlled Trial
Brief Title: Effects of Hip Bump Manipulation Versus Sham Treatment in Healthy Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dominican University New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2025-0328-01
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Assessment of Hip Strength, Range of Motion, EMG Activation, and Landing Mechanics in Healthy Subjects; Healthy Adult Subjects
Keywords: Hip Bump Manipulation; Unrestrained Femoral Internal Rotation; UFIR; HVLAT
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Two-Arm Parallel Group Randomized Controlled Trial (RCT) Group A: Intervention Group B: Control (Sham)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Intervention (Experimental): Hip Bump Manipulation (UFIR)
  Interventions: Procedure: Hip Bump Manipulation
- Group B: Control (Sham Comparator): Iliac Crest Bump Sham Manipulation
  Interventions: Procedure: Sham (No Treatment)

INTERVENTIONS:
Procedure: Hip Bump Manipulation — This technique is a high velocity low amplitude thrust (HVLAT) directly posterior to the greater trochanter which theorizes the quick stretch of the external rotator muscles and may improve a malpositioned femoral head within the acetabulum.
  Other Names: UFIR; Unrestrained Femoral Internal Rotation
  Arms: Group A: Intervention
Procedure: Sham (No Treatment) — Iliac Crest Sham Manipulation
  Arms: Group B: Control

SUMMARY:
The purpose of this study is to objectively assess the effects of hip bump manipulation (HBM) on a healthy population aged 18-45 years. We hypothesize that the HBM will improve hip internal rotation passive range of motion, improve the strength of the hip external rotators, decrease compensatory motions in hip flexion during active range of motion, and improve bipodal landing mechanics.

Human participants will be analyzed to determine whether the manipulation produces the intended clinical outcomes. While clinicians commonly use this technique, its effectiveness has yet to be substantiated through research. This technique is a high velocity low amplitude thrust to the greater trochanter which theorizes the quick stretch of the external rotator muscles and may improve a malpositioned femoral head within the acetabulum. These improvements may positively affect functional movements such as bipodal landing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Aged 18-45 years old

Exclusion Criteria:

* Diagnosed demoroacetabular labral tear
* Diagnosed osteoarthritis (OA)
* Current or recent (within the past 6 months) low back pain
* Hip or pelvic pain
* Lower extremity injury within the past six months
* Diagnosed scoliosis
* History of surgery involving the femoroacetabular joint (FAJ)
* Known allergic reaction to adhesive or shaving cream used for EMG placement

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Hip External Rotation Strength | "From pre-intervention to post-intervention within a single session lasting approximately 20 minutes."
  Measured with ActivForce Handheld Dynamometry. 3 trials for an average Mean Voluntary Isometric Contraction
Hip Internal Rotation Range of Motion | "From pre-intervention to post-intervention within a single session lasting approximately 20 minutes."
  Hip Internal rotation measured in a seat position 90/90 position. Measured with IPhone Digital Goniometry. 3 trials with a calculated average
Hip EMG Muscle Activation | "From pre-intervention to post-intervention within a single session lasting approximately 20 minutes."
  Delsys Trigno Wireless System will be used to monitor changes in muscle activation between the Tensor Fascia Latae, Gluteus Medius, and Gluteus Maximus. During seated isometric external rotation contraction and bipodal landing. EMG will be retrieved on the 2nd attempt out of 3 trials.
Bipodal Landing | "From pre-intervention to post-intervention within a single session lasting approximately 20 minutes."
  Kinvent K-Delta Force Plates used to measure changes in bipodal landing mechanics including force distribution, time to stabilization, etc. 3 trials will be conducted to present average values

SECONDARY OUTCOMES:
Hip Deviation with Active Assisted Hip Flexion Range of Motion | "From pre-intervention to post-intervention within a single session lasting approximately 20 minutes."
  Deviation resulting in excessive abduction and external rotation during knee to chest active assisted range of motion. Video recording before and after to observe changes pre and post intervention.
Hip External Rotation Range of Motion | "From pre-intervention to post-intervention within a single session lasting approximately 20 minutes."
  Measured to compare the change in External and Internal Rotation range of motion relationship. Measure with iPhone Digital Goniometry. 3 trials will be conducted to present an average value of ROM

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Edeer, B.S., M.S., Ph.D., Study Chair — Dominican University New York
Locations (1):
- Dominican University New York, Orangeburg, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data, including demographic information and outcome measures, will be made publicly available as part of the research publication. All personal identifiers will be removed, and any video recordings of movement deviations will either not be shared or will have faces obscured to maintain participant privacy. Data will be provided in a format consistent with ethical guidelines and institutional requirements.

REFERENCES:
- [Background] van Melick N, Meddeler BM, Hoogeboom TJ, Nijhuis-van der Sanden MWG, van Cingel REH. How to determine leg dominance: The agreement between self-reported and observed performance in healthy adults. PLoS One. 2017 Dec 29;12(12):e0189876. doi: 10.1371/journal.pone.0189876. eCollection 2017. PMID 29287067
- [Background] Kazemi M, Leguard SH, Lilja S, Mahaise S. A clinical crossover trial of the effect of manipulative therapy on pain and passive and active range of motion of the painful hip. J Can Chiropr Assoc. 2021 Dec;65(3):318-329. PMID 35197646
- [Background] Bazett-Jones DM, Tylinksi T, Krstic J, Stromquist A, Sparks J. PEAK HIP MUSCLE TORQUE MEASUREMENTS ARE INFLUENCED BY SAGITTAL PLANE HIP POSITION. Int J Sports Phys Ther. 2017 Aug;12(4):535-542. PMID 28900559
- See also: Related Info — https://doi.org/10.1186/s12891-024-07463-5
- See also: Related Info — https://doi.org/10.55225/hppa.548
- See also: Related Info — https://doi.org/10.26603/001c.35577
- See also: Related Info — https://www.ncbi.nlm.nih.gov/books/NBK574527/
- See also: Related Info — https://doi.org/10.26603/001c.89261
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC5638457/
- See also: Related Info — https://doi.org/10.1016/j.jelekin.2020.102457
- See also: Related Info — https://doi.org/10.1371/journal.pone.0189876
- See also: Related Info — https://scholars.indianastate.edu/clinat/vol7/iss3/33/
- See also: Related Info — https://journals.humankinetics.com/view/journals/jsr/32/7/article-p810.xml
- See also: Related Info — https://doi.org/10.1016/j.math.2016.10.013
- See also: Related Info — https://doi.org/10.1371/journal.pone.0230841